CLINICAL TRIAL: NCT01627340
Title: An Open-label Study to Assess the Immunogenicity and Safety of GSK Biologicals' Hepatitis B Vaccine, Engerix™-B in Adults With or Without Type 2 Diabetes Mellitus
Brief Title: Immunogenicity and Safety Study of GlaxoSmithKline (GSK) Biologicals' Engerix™-B in Adults With or Without Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 115918
Record Dates: First submitted 2012-06-21; First posted 2012-06-25 (Estimated); Results first posted 2015-01-09 (Estimated); Last update posted 2018-07-31 (Actual); Status verified 2017-01

CONDITIONS: Hepatitis B
Keywords: Engerix™-B; hepatitis B; adults; Type 2 diabetes mellitus
MeSH Terms: conditions — Hepatitis B; Diabetes Mellitus, Type 2

ARMS (2):
- Diabetes Group (Experimental): Subjects diagnosed with type 2 diabetes within the five year period before study start who received 3 doses of Engerix™-B vaccine (HBV) at 0, 1 and 6 months. The vaccine was administered intramuscularly (IM) into the deltoid region of the non-dominant arm.
  Interventions: Biological: Engerix™-B vaccine
- Control Group (Active Comparator): Subjects with no diagnosis or documented history of diabetes who received 3 doses of Engerix™-B (HBV) vaccine at 0, 1 and 6 months. The vaccine was administered intramuscularly into the deltoid region of the non-dominant arm.
  Interventions: Biological: Engerix™-B vaccine

INTERVENTIONS:
Biological: Engerix™-B vaccine — 3 doses administered intramuscularly (IM) in the deltoid region of the non-dominant arm.
  Other Names: HBV

SUMMARY:
This study will evaluate the immunogenicity and safety of Engerix™-B (hepatitis B vaccine) when administered as a primary vaccination course at 0, 1 and 6 months in adults with or without type 2 diabetes mellitus.

ELIGIBILITY:
Inclusion Criteria:

All subjects must satisfy ALL the following criteria at study entry:

* Subjects who, in the opinion of the investigator, can and will comply with the requirements of the protocol.
* A male or female subject aged 20 years and above at the time of screening.
* Written informed consent obtained from the subject at screening.
* Subjects diagnosed with type 2 diabetes documented within the past five years, according to the criteria specified by the American Diabetes Association or currently taking any form of anti-diabetic intervention documented by the investigator; or control subjects with no diagnosis or documented history of diabetes, and HbA1c less than 6.5%, as determined by laboratory screening tests.
* Normal renal function defined as estimated glomerular filtration rate (GFR) ≥ 50 mL/min, estimated through the Modification of Diet in Renal Disease (MDRD) or the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation, as determined by laboratory screening tests.
* Seronegative for hepatitis B surface antigen (HBsAg), anti-HBs antibodies and antibodies to hepatitis B core antigen (anti HBc), as determined by laboratory screening tests.
* Female subjects of non-childbearing potential may be enrolled in the study.

  * Non-childbearing potential is defined as pre-menarche, current tubal ligation, hysterectomy, ovariectomy or post-menopause.
* Female subjects of childbearing potential may be enrolled in the study, if the subject:

  * has practiced adequate contraception for 30 days prior to vaccination, and
  * has a negative pregnancy test on the day of screening and at Visit 1, and
  * has agreed to continue adequate contraception during the entire treatment period and for two months after completion of the vaccination series.

Exclusion Criteria:

The following criteria should be checked at the time of study entry. If ANY exclusion criterion applies, the subject must not be included in the study:

* Use of any investigational or non-registered product other than the study vaccine within 30 days preceding the first dose of study vaccine, or planned use during the study period.
* Chronic administration of immunosuppressants or other immune-modifying drugs within six months prior to the first vaccine dose.
* Administration of long-acting immune-modifying drugs within 6 months of the study entry or planned administration at any time during the study period.
* Administration of a vaccine not foreseen by the study protocol starting from 30 days before each dose of vaccine and ending 30 days after each dose, with the exception of the inactivated influenza vaccine which is allowed at any time during the study if administered at a separate site.
* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a protocol-specified non-investigational product.
* Any previous complete or incomplete vaccination against hepatitis B since birth.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, including HIV infection, based on medical history and physical examination.
* History of any reaction or hypersensitivity likely to be exacerbated by any component of the vaccine, including latex.
* Advanced heart failure or any other severe clinical condition that significantly reduces the subject's life expectancy.
* Acute disease and/or fever at the time of enrolment.
* Administration of immunoglobulins and/or any blood products within the three months preceding the first dose of study vaccine or planned administration during the study period.
* Any history of alcohol or drug abuse in the past 5 years.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 667 (Actual)
Dates: Start 2012-07-24; Primary Completion 2013-12-18 (Actual); Study Completion 2013-12-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (22):
- United States (10):
  - GSK Investigational Site, Huntsville, Alabama
  - GSK Investigational Site, Stockbridge, Georgia
  - GSK Investigational Site, Boise, Idaho
  - GSK Investigational Site, Mishawaka, Indiana
  - GSK Investigational Site, Wichita, Kansas
  - GSK Investigational Site, Endwell, New York
  - GSK Investigational Site, Cleveland, Ohio
  - GSK Investigational Site, Nashville, Tennessee
  - GSK Investigational Site, Salt Lake City, Utah
  - GSK Investigational Site, Wenatchee, Washington
- Australia (3):
  - GSK Investigational Site, Herston, Queensland
  - GSK Investigational Site, Box Hill, Victoria
  - GSK Investigational Site, St Albans, Victoria
- Canada (5):
  - GSK Investigational Site, Truro, Nova Scotia
  - GSK Investigational Site, Greater Sudbury, Ontario
  - GSK Investigational Site, Kitchener, Ontario
  - GSK Investigational Site, Québec, Quebec
  - GSK Investigational Site, Ste-Foy, Quebec
- New Zealand (4):
  - GSK Investigational Site, Hamilton
  - GSK Investigational Site, Rotorua
  - GSK Investigational Site, Takapuna Auckland
  - GSK Investigational Site, Wellington

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Van Der Meeren O, Peterson JT, Dionne M, Beasley R, Ebeling PR, Ferguson M, Nissen MD, Rheault P, Simpson RW, De Ridder M, Crasta PD, Miller JM, Trofa AF. Prospective clinical trial of hepatitis B vaccination in adults with and without type-2 diabetes mellitus. Hum Vaccin Immunother. 2016 Aug 2;12(8):2197-2203. doi: 10.1080/21645515.2016.1164362. Epub 2016 Apr 28. PMID 27123743
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Statistical Analysis Plan: 115918 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 115918 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 115918 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 115918 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 115918 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 115918 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: There was re-allocation of 7 subjects conducted due to certain discrepancies between subjects' attributes identified from two different sources and as a result of which, there was an increase in the number of subjects from the 667 subjects targeted initially.
Period: Overall Study
Arm/Group | Diabetes Group | Control Group
Started | 416 | 258
Completed | 404 | 254
Not Completed | 12 | 4
Not completed — Adverse Event | 1 | 0
Not completed — Lost to Follow-up | 8 | 4
Not completed — Pregnancy | 1 | 0
Not completed — Withdrawal by Subject | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Diabetes Group | Control Group | Total
Number analyzed (Participants) | 416 | 258 | 674
Age, Continuous [Mean (Standard Deviation); unit: Years] | 53.2 (12.32) | 49.6 (13.72) | 51.8 (12.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 182 | 152 | 334
  Male | 234 | 106 | 340

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Seroprotected for Anti- Hepatitis B Surface Antigen (Anti-HBs) Antibodies
Description: A seroprotected subject was defined as a vaccinated subject with an anti-HBs antibody concentration greater than or equal to (≥) 10 milli-international units per milliliter (mIU/mL).
Time Frame: At one month after the third dose of primary vaccination (Month 7)
Population: The analysis was performed on the According-to-Protocol (ATP) cohort for immunogenicity, which included all evaluable subjects who received all 3 doses of the EngerixTM-B vaccine, for whom post-vaccination immunogenicity results were available and for those in the Control Group, a suitable match was available in the Diabetic Group.
Measure: Count of Participants; unit: Participants
Arm/Group | Diabetes Group | Control Group
Number analyzed (Participants) | 378 | 189
Participants | 285 | 155

2. Secondary Outcome: Anti-HBs Antibody Concentration
Description: Concentrations were given as geometric mean concentration (GMC) and expressed as mIU/mL
Time Frame: At one month after the third dose of primary vaccination (Month 7)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | Diabetes Group | Control Group
Number analyzed (Participants) | 378 | 189
mIU/mL | 147.6 [110.2 to 197.8] | 384.2 [254.5 to 580.0]

3. Secondary Outcome: Number of Subjects Reporting Any Solicited Local Symptoms
Description: Solicited local symptoms assessed were pain, redness and swelling. Any was defined as occurrence of the specified solicited local symptom regardless of its intensity grade.
Time Frame: During the 4-day (Days 0-3) post-vaccination period
Population: The analysis was performed on Total Vaccinated cohort, which included all subjects who received at least one study vaccine administration and had symptom sheet completed.
Measure: Count of Participants; unit: Participants
Arm/Group | Diabetes Group | Control Group
Number analyzed (Participants) | 413 | 257
Participants
  Any Pain | 160 | 115
  Any Redness | 84 | 51
  Any Swelling | 49 | 19

4. Secondary Outcome: Number of Subjects Reporting Any Solicited General Symptoms
Description: Solicited general symptoms assessed were fatigue, gastrointestinal symptoms, headache and fever. Any was defined as any solicited general symptom reported irrespective of intensity and relationship to vaccination. Any fever = oral temperature greater than or equal to (≥) 37.5 degrees Celsius (°C)
Time Frame: During the 4-day (Days 0-3) post-vaccination period
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Diabetes Group | Control Group
Number analyzed (Participants) | 413 | 257
Participants
  Any Fatigue | 118 | 69
  Any Gastrointestinal symptoms | 83 | 47
  Any Headache | 97 | 71
  Any Fever | 15 | 8

5. Secondary Outcome: Number of Subjects Reporting Any Unsolicited Adverse Events (AEs)
Description: An unsolicited AE was defined as an untoward medical occurrence in a patient or clinical investigation subject, temporally associated with use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as occurrence of any unsolicited symptom regardless of intensity grade or relation to vaccination.
Time Frame: During the 31-day (Days 0-30) post-vaccination period
Population: The analysis was performed on the Total Vaccinated cohort, which included all subjects who received at least one study vaccine administration.
Measure: Count of Participants; unit: Participants
Arm/Group | Diabetes Group | Control Group
Number analyzed (Participants) | 416 | 258
Participants | 150 | 96

6. Secondary Outcome: Number of Subjects Reporting Any Serious Adverse Events (SAEs)
Description: A serious adverse event was defined as any untoward medical occurrence that: resulted in death, was life threatening, required hospitalization or prolongation of hospitalization, resulted in disability/incapacity or was a congenital anomaly/birth defect in the offspring of a study subject. Any was defined as occurrence of any symptom regardless of intensity grade or relation to vaccination.
Time Frame: During the entire study period (Month 0 - Month 7)
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Groups:
- Diabetes Group: Subjects diagnosed with type 2 diabetes within the five year period before study start who received 3 doses of EngerixTM-B vaccine (HBV) at 0, 1 and 6 months. The vaccine was administered intramuscularly (IM) into the deltoid region of the non-dominant arm.
- Control Group: Subjects with no diagnosis or documented history of diabetes who received 3 doses of EngerixTM-B (HBV) vaccine at 0, 1 and 6 months. The vaccine was administered intramuscularly into the deltoid region of the non-dominant arm.
Arm/Group | Diabetes Group | Control Group
Number analyzed (Participants) | 416 | 258
Participants | 16 | 4

ADVERSE EVENTS:
Time Frame: Serious Adverse Events: From Month 0 to Month 7; Solicited local and general symptoms: During the 4-day (Days 0-3) post-vaccination period.
Description: For the systematically assessed other (non-serious) adverse events, the number of participants at risk included those from Total Vaccinated Cohort who had the symptom sheet completed.
Arm/Group | Diabetes Group | Control Group
Serious Adverse Events (participants affected / at risk) | 16/416 | 4/258
Other Adverse Events (participants affected / at risk) | 247/416 | 168/258
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Diabetes Group (N=416) | Control Group (N=258)
Dehydration (Metabolism and nutrition disorders) | 1 | 1
Anaphylactic reaction (Immune system disorders) | 1 | 0
Angina unstable (Cardiac disorders) | 1 | 0
Appendicitis (Infections and infestations) | 1 | 0
Brain neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Concussion (Injury, poisoning and procedural complications) | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 1
Glioblastoma multiforme (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Incisional hernia, obstructive (Injury, poisoning and procedural complications) | 1 | 0
Infected skin ulcer (Infections and infestations) | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1
Mediastinitis (Infections and infestations) | 0 | 1
Mitral valve disease (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 1 | 0
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Oedema peripheral (General disorders) | 1 | 0
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pelvic inflammatory disease (Infections and infestations) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Radius fracture (Injury, poisoning and procedural complications) | 1 | 0
Renal failure (Renal and urinary disorders) | 1 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0
Scapula fracture (Injury, poisoning and procedural complications) | 1 | 0
Syncope (Nervous system disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Diabetes Group (N=416) | Control Group (N=258)
Pain (General disorders) | 160 | 115
Redness (General disorders) | 84 | 51
Swelling (General disorders) | 49 | 19
Fatigue (General disorders) | 118 | 69
Gastrointestinal symptoms (General disorders) | 83 | 47
Headache (General disorders) | 97 | 71

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.